CLINICAL TRIAL: NCT02149914
Title: The Changes of Ryodoraku and HRV After PPI Treatment in GERD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Mei-Ling Shen, Mei-Ling Shen, Taichung Tzu Chi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: REC103-20
Record Dates: First submitted 2014-05-18; First posted 2014-05-29 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Non-erosive Reflux Disease; Barrett's Esophagus
Keywords: Ryodoraku; Meridian energy; Heart rate variability; Autonomic Nervous System; GERD
MeSH Terms: conditions — Non-Erosive Reflux Disease; Barrett Esophagus; Gastroesophageal Reflux | interventions — Proton Pump Inhibitors; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PPI treatment (Experimental): Patients with GERD would be assessed by ANSWatch. Ryodoraku, UGI endoscopy, and GerdQ before taking PPIs and after taking PPI 20mg tablet by mouth everyday for 4 weeks.
  Interventions: Device: Ryodoraku; Device: ANSWatch; Device: UGI endoscopy; Other: GerdQ; Drug: PPI

INTERVENTIONS:
Device: Ryodoraku — Ryodoraku to assess the energy of meridian system for each patient before and after taking the medication
  Other Names: Meridian energy analysis device; M.E.A.D; Skin Response Measurement Device; Me-Professional; Me-100
Device: ANSWatch — ANSWatch to assess the autonomic nervous system for each patient before and after taking the medication
  Other Names: "Taiwan Scientific" Noninvasive Blood Pressure Meter; Wrist-worn heart rate monitor; TS-0411
Device: UGI endoscopy — UGI endoscopy to assess the grade of reflux esophagitis for each patient before and after taking the medication
  Other Names: Upper gastrointestinal endoscope; Fujinon EG350N; Fujinon EG590WR
Other: GerdQ — GerdQ to assess the severity of GERD for each patient before and after taking the medication
  Other Names: Gastroesophageal reflux disease questionnaire
Drug: PPI
  Other Names: Proton Pump Inhibitor; Rabeprazole; Pariet

SUMMARY:
Gastroesophageal reflux disease(GERD) mainly related to the reflux of stomach content induced by the dysfunction of lower esophageal sphincter. Proton pump inhibitors (PPI) can effectively block gastric acid secretion but the drug reactions and the degree of improvement in symptoms are sometimes unpredictable. The aim of this study is to investigate the association between the clinical efficacy of PPI in patients with GERD and the personal physical status by Ryodoraku and ANSWatch.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease(GERD) is a common disease, mainly related to the reflux of stomach content induced by the dysfunction of lower esophageal sphincter. The common symptoms of GERD are heartburn, acid regurgitation, chest pain and globus hystericus. The methods to treat GERD are changes of lifestyle, pharmacotherapy, antireflux surgery and endoscopy. Proton pump inhibitors (PPI) can effectively block gastric acid secretion and promote the repair of esophagus, but the drug reactions and the degree of improvement in symptoms are sometimes unpredictable. Recently there are many instruments used to analyze personal physical status. Meridian energy analysis device ( Ryodoraku ) is used to assess the energy of meridian system by analysis of resistance of the skin surface, as well as the wrist-worn heart rate monitor (ANSWatch) used to assess the autonomic nervous system by analysis of heart rate variability. Therefore, the aim of this study is to investigate the association between the clinical efficacy of PPI in patients with GERD and the personal physical status by Ryodoraku and ANSWatch.

Investigators will recruit 120 patients with GERD in clinic who have to receive PPIs for four weeks and assess each volunteer before and after taking the medication. Assessment methods : 1. ANSWatch to assess the autonomic nervous system, 2. Ryodoraku to assess the energy of meridian system, 3. Upper gastrointestinal endoscopy to assess the grade of reflux esophagitis, 4. gastroesophageal reflux disease questionnaire to assess the severity of GERD. Investigators analysed and compared the database from the assessments between before and after taking the medication.

Investigators anticipate to substantiate that the changes of Ryodoraku and ANSWatch are good predictors for the clinical efficacy of PPI in patients with GERD.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age of 20-75 years
* patients with GERD who have to receive PPIs for four weeks

Exclusion Criteria:

* Suffering from peptic ulcer, gallstones, cancer, and Barrett's esophagus
* previously underwent the esophagus, stomach or duodenum surgery
* Lactating women or pregnant women

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
gastroesophageal reflux disease questionnaire | four weeks
  To assess the severity of GERD

SECONDARY OUTCOMES:
Upper gastrointestinal endoscopy | four weeks
  To assess the grade of reflux esophagitis

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Ling Shen, M.D, Study Chair — Taichung Tzu Chi Hospital
Locations (1):
- Taichung Tzu Chi Hospital, Taichung, Taiwan, Taiwan